CLINICAL TRIAL: NCT05383014
Title: Assessment of Association Between FLT3-ITD Gene Mutation and CD135 Expression and Their Correlation With Hematological,Immunophenotypic and Biochemical Characteristics in Acute Myeloid Leukemia.
Brief Title: FLT3-ITD Gene Mutation and CD135 Expression in Acute Myeloid Leukemia.
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Shaimaa Abd Elazeem Saber Selim, Assist. lecturer, Assiut University
Other Study IDs: FLT3-ITD and CD135 in AML
Record Dates: First submitted 2022-05-17; First posted 2022-05-19 (Actual); Last update posted 2022-05-19 (Actual); Status verified 2022-05

CONDITIONS: Acute Myeloid Leukemia
MeSH Terms: conditions — Leukemia, Myeloid, Acute

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — FLT3-ITD mutations will be determined from genomic DNA using polymerase chain reaction (PCR)-based method on Peripheral blood samples of AML patients
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
1. To evaluate expression levels of CD135
2. To assess the frequency of FLT3 gene mutations (ITD)
3. association between FLT3-ITD mutation and CD135 expression and their correlation with hematological, immunophenotypic,and biochemical features.

DETAILED DESCRIPTION:
Acute leukemias are clonal malignant diseases of immature hematopoietic system ,characterized by clonal evolution and considerable genetic, epigenetic, and phenotypic heterogeneity,and constitute a common cause of morbidity and mortality worldwide.[1] Gene expression profiling has improved the molecular classification and prognosis of Acute leukemias, where molecular testing has become mandatory for further classify into prognostic groups. Among the genetic aberrations, alterations of the FMS-like tyrosine kinase 3 (FLT3) gene. [2] FLT3 is a type 3 receptor tyrosine kinase that plays an important role in the expansion and proliferation of multi-potent progenitor cells within the bone marrow.[3] mutations of FLT3 induce a constitutional activation of tyrosine kinases and several downstream targets resulting in proliferation and growth of malignant cells ,myeloproliferative phenotype , high tumor burden,and a characteristic hematological , immunophenotypic and biochemical profile that can be identified during routine diagnostic workup.[4]Two mutations exist in these cells: FLT3-ITD (internal tandem duplication), and FLT3-TKD, a point mutation in the tyrosine kinase domain.[5] FLT3-ITD is a common driver mutation, seen with a frequency of 20 to 30% ,and significantly affecting the pathogenesis and the clinical outcome . Genetic testing for FLT3-ITD mutation at diagnosis is done to risk stratify patients and to guide therapeutic decisions.[6-8] FLT3 receptor/CD135 is a transmembrane tyrosine kinase receptor, normally expressed on the surface of hematopoietic stem cells and is lost upon cell differentiation , activation of the receptor resulting in stimulating survival and proliferation, and inhibiting apoptosis of progenitor cells . Overexpression of the FLT3 receptor has been reported to be associated with high risk for relapse in patients with acute leukemia .[2]

ELIGIBILITY:
Inclusion Criteria:

* Newly diagnosed Patients with acute myeloid leukemia (AML), who fullfill the WHO criteria.

Exclusion Criteria:

* AML on top of myeloproliferative neoplasms or MDS.
* previously diagnosed AML on treatment
* Patients with any other type of malignant tumors

Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: Newly diagnosed Patients with acute myeloid leukemia (AML), who fullfill the WHO criteria.
Sampling Method: Non-Probability Sample
Enrollment: 82 (Estimated)
Dates: Start 2022-06-01 (Estimated); Primary Completion 2024-06-01 (Estimated); Study Completion 2024-07-01 (Estimated)

PRIMARY OUTCOMES:
Correlation between FLT3 gene mutation and the expression of CD135 and their association with clinical outcome ,haematological, immunophenotypic , biochemical characteristics in the development and progression of AML. | baseline
  analysis of association between FLT3 gene mutation and the level of expression of CD135 and analysis of clinical outcome , hematological,and immunophenotypic characteristics between patients with positive FLT3-ITD mutation and negatine patients

SECONDARY OUTCOMES:
To detect expression levels of CD135 and the frequency of FLT3- ITD gene mutations in the development and progression of AML -follow up of patient after induction of chemotherapy | baseline

CONTACTS AND LOCATIONS:
Overall Officials: Marwa Mohammed Thabet, lecturer, Study Director — clinical pathology department , Assiut University Hospital.; Alaa soliman Abd Elkadir, lecturer, Study Director — clinical pathology department , Assiut University Hospital.

REFERENCES:
- [Background] Vela-Ojeda J, Cardenas PV, Garcia-Ruiz Esparza MA, Montiel Cervantes LA, Chavez JG, Caballero AH, Majluf-Cruz A, Vega-Lopez A, Reyes-Maldonado E. FLT3-ITD and CD135 Over-Expression are Frequent Findings of Poor Survival in Adult Patients with Acute Leukemias. Arch Med Res. 2021 Feb;52(2):217-223. doi: 10.1016/j.arcmed.2020.10.013. Epub 2020 Oct 24. PMID 33109387
- [Background] Ambinder AJ, Levis M. Potential targeting of FLT3 acute myeloid leukemia. Haematologica. 2021 Mar 1;106(3):671-681. doi: 10.3324/haematol.2019.240754. PMID 32703795
- [Background] Gilliland DG, Griffin JD. The roles of FLT3 in hematopoiesis and leukemia. Blood. 2002 Sep 1;100(5):1532-42. doi: 10.1182/blood-2002-02-0492. PMID 12176867
- [Background] Juliusson G, Jadersten M, Deneberg S, Lehmann S, Mollgard L, Wennstrom L, Antunovic P, Cammenga J, Lorenz F, Olander E, Lazarevic VL, Hoglund M. The prognostic impact of FLT3-ITD and NPM1 mutation in adult AML is age-dependent in the population-based setting. Blood Adv. 2020 Mar 24;4(6):1094-1101. doi: 10.1182/bloodadvances.2019001335. PMID 32203582
- [Background] Daver N, Schlenk RF, Russell NH, Levis MJ. Targeting FLT3 mutations in AML: review of current knowledge and evidence. Leukemia. 2019 Feb;33(2):299-312. doi: 10.1038/s41375-018-0357-9. Epub 2019 Jan 16. PMID 30651634
- [Background] Khera R, Ahmed F, Mundada M, Nambaru L, Murthy SS, Devig S, Rajappa SJ, Mallavarapu KM, Santa A, Kumar P. Acute Myeloid Leukaemia with Gene Mutation: A Correlation with Haematological and Immunophenotypic Characteristics and Our Experience in a Tertiary Care Cancer Center in South India. Turk Patoloji Derg. 2018;34(2):171-174. doi: 10.5146/tjpath.2017.01415. PMID 28984348